CLINICAL TRIAL: NCT05861388
Title: Short Term Comparative Evaluation of Bio-HPP and Cast Cobalt-chromium as a Framework for Implant-supported Prostheses: A Split-mouth Clinical Randomized Study
Brief Title: Bio-HPP vs Cast Co-cr as Implant Framework
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Mohammed Amer, assistant lecturer at prosthodontic department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prosth16/06/02
Record Dates: First submitted 2021-10-20; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Bio-HPP; PEEK; Screw-Retained; Implant Framework

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cobalt chrome implant framework (Active Comparator): the participants received Co-Cr based screw-retained implant supported prosthesis at one side of the lower jaw
  Interventions: Procedure: implant placement
- Bio-Hpp implant framework (Experimental): The participants received Bio-Hpp based screw-retained implant-supported prosthesis at the other side
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — 2 implants were placed at position of lower 2nd premolar and 2nd molar
  Other Names: final prosthesis was constructed on the implants

SUMMARY:
The purpose of this study was to assess the effect of Bio-Hpp versus Co-Cr custom abutments in fixed-detachable implant-supported mandibular partial dentures clinically and radiographically in Class I Kennedy classification (split-mouth study)

DETAILED DESCRIPTION:
Participants with bilateral partial edentulism in the posterior mandible received two implants at the positions of the second premolar and second molar on both sides; one side was restored with BioHpp based screw-retained FDP (test group) and the other side was restored with Co-Cr based screw-retained FDP (control group). All patients were clinically examined at the time of prosthesis insertion, and 6,12 months later for fracture of implant or framework, fracture, or looseness of the screw, veneer chipping, and fractures, modified bleeding index, modified plaque index, peri-implant probing depth, as well as radiographically for marginal bone loss

ELIGIBILITY:
Inclusion Criteria:

* Mandibular posterior edentulous with the first premolar as the last standing abutment tooth bilaterally.

  * All patients were edentulous for at least 6 months from the last extraction.
  * The bone height of the alveolar ridge was not less than 12 mm above the inferior alveolar canal and the buccolingual width of the alveolar ridge at the prospective implant site was not less than 6 mm.
  * The opposing arch was almost dentulous, and any missing teeth were restored using a fixed partial denture.
  * Adequate interarch space at least 5mm between the opposing dentition and the mandibular edentulous space.
  * Remaining teeth were in good periodontal condition.
  * Maintaining good oral hygiene and were ready to cooperate throughout the study.

Exclusion Criteria:

* Patients with active infection or inflammation or flabby tissue in the areas intended for implant placement.

  * Those patients with systemic diseases that may influence soft or hard tissue healing.
  * Patients with a history of radiation therapy in the head and neck region.
  * Neurological or psychiatric handicap patients that could interfere with good oral hygiene.
  * Heavy smokers and drug abusers.
  * Patients with severe clenching or bruxism.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
marginal bone loss around implants | 12 months
  Marginal bone level was measured from the implant shoulder to the first bone to implant contact on the mesial and distal sides of the implant on digital standardized periapical radiograph using the long cone paralleling technique
modified plaque index | 12 months
  Plaque adherent to the implants was quantified at four surfaces: buccal, lingual, mesial, and distal using a plastic periodontal probe after air drying for the implant and gingiva. The four sides for each implant were scored 0-3 according to the following criteria:
  Score 0: No plaque detected. Score 1: Plaque can be detected by running a probe across the marginal surface of the implant.
  Score 2: Plaque can be seen by naked eye. Score 3: Abundance of plaque.
modified bleeding index | 12 months
  A plastic periodontal probe was passed along the gingival margin adjacent to the implant and the following scores were given according to Mombelli and Lang Score 0: No bleeding with slight pressure on the mucosa using periodontal probe.
  Score 1: Isolated bleeding spots visible. Score 2: Blood forms a confluent red line on margin. Score 3: Heavy or profuse bleeding
probing depth | 12 months
  ., the peri- implant probing pocket depth is measured around the surfaces of the implants in four areas (mid-buccal, mid-lingual, med-mesial, mid-distal) using plastic periodontal probe* which was inserted with light force and parallel to long axis of implant

SECONDARY OUTCOMES:
mechanical complications | 12 months after loading
  framework fracture, screw loosening, screw fracture and chipping or fracture of veneer layer

IPD SHARING:
Plan to Share IPD: No